CLINICAL TRIAL: NCT05448664
Title: Health Belief Model and Family-based Mobile-health Intervention to Promote Oral Health in Adolescents: A Cluster Randomized Controlled Trial
Brief Title: Mobile-health Intervention to Promote Oral Health in Adolescents: A Cluster Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr Liu, Pei Pearl, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HMRF 19201281
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Oral Health
Keywords: Mobile health; Health Belief Model; Family-based intervention; Oral health; Adolescents

STUDY DESIGN:
Intervention Model Description: Three-arm parallel design cluster randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Families HBM- mobile messaging (Experimental): Family- and HBM-based behavioral intervention using mobile messaging
  Interventions: Behavioral: Family HBM- mobile messaging
- Adolescents HBM- mobile messaging (Active Comparator): Student- and HBM-based behavioral intervention using mobile messaging
  Interventions: Behavioral: Adolescent HBM- mobile messaging
- Adolescents e-pamphlets (Placebo Comparator): Prevailing oral health education by e-version of pamphlets through mobile messaging
  Interventions: Behavioral: Adolescent e-pamphlets

INTERVENTIONS:
Behavioral: Family HBM- mobile messaging — The intervention will consist of two blocks of text messaging based on HBM model, the messages will be sent to the students and their parents in the following 24 weeks.
  Arms: Families HBM- mobile messaging
Behavioral: Adolescent HBM- mobile messaging — The intervention will consist of two blocks of text messaging based on HBM model, the messages will be sent to the students in the following 24 weeks.
  Arms: Adolescents HBM- mobile messaging
Behavioral: Adolescent e-pamphlets — The contents of e-version of three pamphlets, published by Department of Health (http://www.toothclub.gov.hk/en/en_index.html) will be distributed in an electronic form and sent via a mobile message.
  Arms: Adolescents e-pamphlets

SUMMARY:
The aim of this study is to investigate the effectiveness of the family and behavioral theory based mobile-health behavioral intervention in enhancing adolescents'good oral health behaviors (mainly oral hygiene practice and free sugar intake control) and preventing common oral diseases (dental caries and periodontal diseases).

DETAILED DESCRIPTION:
The investigators propose a 30-months clustered randomized controlled trial to investigate the effectiveness of Health Belief Model (HBM) and family-based mobile-health intervention in enhancing the adolescents' good oral health behaviors and preventing oral diseases.

This is a three-arm parallel-design cluster-randomized controlled trial. Parents and their children (12 to 15-year-old) will be recruited and randomized into 3 groups based on the school sites.

Messages targeted on six domains guided by HBM will be sent to the adolescents and their parents via mobile phone. Two blocks of HBM-based oral health messages, reminders, feedback and reinforcement messages will be delivered to both students and parents by mobile phone for 24 weeks; while the intervention of the other 2 groups will target on students only or using prevailing oral health education.

The primary outcomes will be caries increment of the adolescents 2-year post-intervention. Change in oral health self-efficacy and behaviors, dental plaque and gingival bleeding index will be the secondary outcomes.

The investigators anticipate the proposed family- and HBM-based behavioral intervention is more effective than HBM-based mobile-health intervention on adolescents alone or prevailing oral health education in improving the adolescents' oral hygiene behaviors, reducing free-sugar intake and preventing oral diseases.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity;
* Student living with their own parent(s) or primary caregivers;
* Both student and parent(s) or primary caregiver having their own access to a personal mobile phone with certain Apps to receive the messages in time

Exclusion Criteria:

* Student currently on a special diet (e.g. severe inflammatory bowel disease);
* Student has medical conditions know to affect growth or eating (e.g. diabetes, cystic fibrosis);
* Enrollment in other oral health promotion programs or research studies.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Caries increment | 2 years
  Dental caries increment (by tooth level) from baseline to 2 years follow up

SECONDARY OUTCOMES:
Change of oral health self-efficacy | 2 years
  Change from baseline self-efficacy at 2 years
Change of gingival status | 2 years
  Change from baseline gingival bleeding (BOP%) at 2 years, as recommended by the WHO for conducting oral health surveys
Change of toothbrushing behavior | 2 years
  Change from baseline average frequency of toothbrushing per day at 2 years
Change of free-sugar intake | 2 years
  Change from baseline average frequency of intake of sugary snack/drink per day at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pei LIU, Principal Investigator — The University of Hong Kong
Locations (1):
- Faculty of Dentistry, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu P, Wong MCM, Lee GHM, Yiu CKY, Lo ECM. Family behavior theory-based intervention via mobile messaging to improve oral health of adolescents: study protocol for a cluster randomized controlled trial. Trials. 2022 Nov 16;23(1):941. doi: 10.1186/s13063-022-06861-1. PMID 36384815